CLINICAL TRIAL: NCT03609814
Title: Population Pharmacokinetics of the Nucleoside Analogues Clofarabine and Fludarabine in Pediatric Patients Undergoing Hematopoietic Cell Transplantation (alloHCT)
Brief Title: Study of Clofarabine and Fludarabine Drug Exposure in Pediatric Bone Marrow Transplantation (HCT)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: P1518454; 19081 (Other: University of California, San Francisco)
Record Dates: First submitted 2018-01-05; First posted 2018-08-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Hematologic Malignancies; Nonmalignant Diseases; Immunodeficiencies; Hemoglobinopathies; Genetic Inborn Errors of Metabolism; Fanconi's Anemia; Thalassemia; Sickle Cell Disease
Keywords: fludarabine; clofarabine; pharmacokinetics; pediatric; allogeneic
MeSH Terms: conditions — Hematologic Neoplasms; Immunologic Deficiency Syndromes; Hemoglobinopathies; Fanconi Anemia; Thalassemia; Anemia, Sickle Cell | interventions — Clofarabine; fludarabine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Bone Marrow Transplantation Recipients: Children undergoing alloHCT at UCSF Benioff Children's Hospital.
  Interventions: Drug: Clofarabine; Drug: Fludarabine Injection

INTERVENTIONS:
Drug: Clofarabine — Given IV
Drug: Fludarabine Injection — Given IV

SUMMARY:
Fludarabine and clofarabine are chemotherapy drugs used extensively in bone marrow transplantation. The goal of this study is to determine what causes some children to have different drug concentrations of clofarabine and fludarabine in their bodies and if drug levels are related to whether or not a child experiences severe side-effects during their bone marrow transplant. The hypothesis is that clinical and individual factors cause changes in clofarabine and fludarabine drug levels in pediatric bone marrow transplant patients and that high levels may cause severe side-effects.

DETAILED DESCRIPTION:
Fludarabine and clofarabine are nucleoside analogs with potent antitumor and immunosuppressive properties used in conditioning regimens of pediatric allogeneic hematopoietic cell transplantation (alloHCT) to promote stem cell engraftment.

This is a single-center, prospective, non-interventional pharmacokinetic (PK) study investigating the clinical pharmacology of combination nucleoside analogue therapy in 24 children undergoing alloHCT at University of California, San Francisco Benioff Children's Hospital.

Patients would receive clofarabine and fludarabine regardless of whether or not they decide to consent to PK sampling.

Clofarabine and fludarabine doses will not be adjusted based on PK data.

The investigators will apply the combination of a limited sampling strategy and population PK methodologies to determine specific factors influencing clofarabine and fludarabine exposure in pediatric alloHCT recipients and identify exposure-response relationships.

Subjects will undergo PK sampling of clofarabine and fludarabine drug concentrations over the duration of combination therapy (3 to 5 days).

To evaluate sources of variability impacting clofarabine and fludarabine exposure clinical data will be obtained from the patient's medical chart on each day of PK sampling.

To assess exposure-response relationships neutrophil engraftment, treatment-related toxicity, and survival data will be collected through day 100 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Children 0-17 years of age
* Undergoing alloHCT for the treatment of malignant or nonmalignant disorder
* Receiving clofarabine and fludarabine-based preparative regimen

Exclusion Criteria:

* Any child 7-17 years of age unwilling to provide assent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target population for the proposed study includes children 0-17 years of age undergoing alloHCT for the treatment of malignant and nonmalignant disorders. Patients receiving clofarabine and fludarabine over 3 to 5 days are eligible to participate. All patients enrolled in this study will undergo PK sampling on the inpatient pediatric BMT unit at UCSF Benioff Children's Hospital. The proposed research will not study any patients receiving clofarabine and fludarabine in a clinic or any other out-patient setting.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine and clofarabine dual therapy for HCT in pediatric patients. | 2hours post start on infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine and clofarabine dual therapy for HCT in pediatric patients. | 3hours post start of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine and clofarabine dual therapy for HCT in pediatric patients. | 6hours post start of infusion
Analysis of the Area under the Plasma Concentration versus Time Curve (AUC) of fludarabine and clofarabine dual therapy for HCT in pediatric patients. | 24hours post start of infusion

SECONDARY OUTCOMES:
Evaluate the event free survival according to the AUC of fludarabine and clofarabine dual therapy | 1month post transplant
Evaluate the event free survival according to the AUC of fludarabine and clofarabine dual therapy | 3 months post transplant
Evaluate the event free survival according to the AUC of fludarabine and clofarabine dual therapy | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Janel Long-Boyle, PharmD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No